CLINICAL TRIAL: NCT06419374
Title: A Phase 3 Study to Evaluate the Efficacy and Safety of Pegozafermin in Subjects With Compensated Cirrhosis Due to Metabolic Dysfunction-Associated Steatohepatitis (MASH) (ENLIGHTEN-Cirrhosis)
Brief Title: A Study to Evaluate the Efficacy and Safety of Pegozafermin in Participants With Compensated Cirrhosis Due to MASH
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: 89bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIO89-100-132
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Metabolic Dysfunction-Associated Steatohepatitis (MASH) / Nonalcoholic Steatohepatitis (NASH) With Compensated Cirrhosis
Keywords: Liver disease; Fatty Liver; Digestive System Diseases; Metabolic diseases; Metabolic Dysfunction-Associated Steatohepatitis; MASH; Nonalcoholic steatohepatitis; NASH; Metabolic dysfunction-associated steatotic liver disease; MASLD; Nonalcoholic fatty liver disease; NAFLD; Fibrosis; Cirrhosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases; Fatty Liver; Digestive System Diseases; Metabolic Diseases; Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pegozafermin (Experimental)
  Interventions: Biological: Pegozafermin
- Placebo (Placebo Comparator): Matched placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Pegozafermin — Subcutaneous injection
  Other Names: BIO89-100
  Arms: Pegozafermin
Drug: Placebo — Subcutaneous injection
  Arms: Placebo

SUMMARY:
The study will assess the efficacy and safety of pegozafermin administered in participants with compensated cirrhosis due to MASH (biopsy-confirmed fibrosis stage F4 MASH [previously known as nonalcoholic steatohepatitis, NASH]).

ELIGIBILITY:
Key Inclusion Criteria:

* Males or non-pregnant females aged between 18 and 75 years (inclusive) at time of signing the informed consent form (ICF).
* Participants must have type 2 diabetes mellitus diagnosed at least 3 months before screening or at least 2 metabolic risk factors.
* Biopsy-confirmed fibrosis stage F4 MASH (NASH Clinical Research Network (CRN) system) with compensated cirrhosis.
* Body mass index (BMI) at screening ≥25.0 (≥23.0 for Asian participants) and <50.0 kilograms (kg)/meters squared (m^2).

Key Exclusion Criteria:

* Liver disorder other than MASH.
* History or evidence of hepatic decompensation.
* History or evidence of hepatocellular carcinoma.
* Have type 1 diabetes mellitus or poorly controlled type 2 diabetes mellitus.
* ALT or aspartate aminotransferase (AST) ≥250 units per liter (U/L).
* Participants taking vitamin E (>400 international units [IU]/day) must be on stable dose for at least 6 months prior to screening.

Other protocol-defined inclusion and exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 762 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2031-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Achieving Fibrosis Regression | Baseline through Month 24
  Fibrosis regression is defined as improvement in fibrosis by ≥1 stage, at Month 24 biopsy relative to baseline biopsy.
Time to First Occurrence of Disease Progression as Measured by Composite of Protocol -Specified Clinical Events | Baseline up to 5 years

SECONDARY OUTCOMES:
Change from Baseline in Enhanced Liver Fibrosis (ELF) Score | Baseline, up to Month 60
Change from Baseline in Alanine Aminotransferase (ALT) Level | Baseline, up to Month 60
Change from Baseline in FibroScan Vibration-controlled Transient Elastography (VCTE) | Baseline, up to Month 60
Proportion of Participants who Develop Clinically Significant Portal Hypertension (CSPH) | Baseline up to Month 60

CONTACTS AND LOCATIONS:
Overall Officials: Maya Margalit, MD, Study Director — 89bio, Inc.
Locations (231):
- United States (109):
  - 89bio Clinical Study Site, Birmingham, Alabama
  - 89bio Clinical Study Site, Homewood, Alabama
  - 89bio Clinical Study Site, Chandler, Arizona
  - 89bio Clinical Study Site, Flagstaff, Arizona
  - 89bio Clinical Study Site, Peoria, Arizona
  - 89bio Clinical Study Site, Phoenix, Arizona
  - 89bio Clinical Study Site, Tucson, Arizona
  - 89bio Clinical Study Site, Little Rock, Arkansas
  - 89bio Clinical Study Site, North Little Rock, Arkansas
  - 89bio Clinical Study Site, Camarillo, California
  - 89bio Clinical Study Site, Canoga Park, California
  - 89bio Clinical Study Site, Coronado, California
  - 89bio Clinical Study Site, Fountain Valley, California
  - 89bio Clinical Study Site, Fresno, California
  - 89bio Clinical Study Site, Huntington Park, California
  - 89bio Clinical Study Site, La Jolla, California
  - 89bio Clinical Study Site, Los Angeles, California
  - 89bio Clinical Study Site, Pasadena, California
  - 89bio Clinical Study Site, Poway, California
  - 89bio Clinical Study Site, Redwood City, California
  - 89bio Clinical Study Site, Rialto, California
  - 89bio Clinical Study Site, Sacramento, California
  - 89bio Clinical Study Site, Santa Ana, California
  - 89bio Clinical Study Site, Littleton, Colorado
  - 89bio Clinical Study Site, Clermont, Florida
  - 89bio Clinical Study Site, Fort Myers, Florida
  - 89bio Clinical Study Site, Gainesville, Florida
  - 89bio Clinical Study Site, Hialeah Gardens, Florida
  - 89bio Clinical Study Site, Homestead, Florida
  - 89bio Clinical Study Site, Jacksonville, Florida
  - 89bio Clinical Study Site, Lady Lake, Florida
  - 89bio Clinical Study Site, Lakewood Rch, Florida
  - 89bio Clinical Study Site, Lehigh Acres, Florida
  - 89bio Clinical Study Site, Maitland, Florida
  - 89bio Clinical Study Site, Miami, Florida
  - 89bio Clinical Study Site, New Port Richey, Florida
  - 89bio Clinical Study Site, Ocala, Florida
  - 89bio Clinical Study Site, Ocoee, Florida
  - 89bio Clinical Study Site, Orlando, Florida
  - 89bio Clinical Study Site, University Park, Florida
  - 89bio Clinical Study Site, Viera, Florida
  - 89bio Clinical Study Site, Winter Park, Florida
  - 89bio Clinical Study Site, Athens, Georgia
  - 89bio Clinical Study Site, Atlanta, Georgia
  - 89bio Clinical Study Site, Chicago, Illinois
  - 89bio Clinical Study Site, Hammond, Indiana
  - 89bio Clinical Study Site, New Albany, Indiana
  - 89bio Clinical Study Site, South Bend, Indiana
  - 89bio Clinical Study Site, Iowa City, Iowa
  - 89bio Clinical Study Site, Kansas City, Kansas
  - 89bio Clinical Study Site, Topeka, Kansas
  - 89bio Clinical Study Site, Lafayette, Louisiana
  - 89bio Clinical Study Site, Baltimore, Maryland
  - 89bio Clinical Study Site, Glen Burnie, Maryland
  - 89bio Clinical Study Site, Greenbelt, Maryland
  - 89bio Clinical Study Site, Burlington, Massachusetts
  - 89bio Clinical Study Site, Ann Arbor, Michigan
  - 89bio Clinical Study Site, Clinton Township, Michigan
  - 89bio Clinical Study Site, Detroit, Michigan
  - 89bio Clinical Study Site, Wyoming, Michigan
  - 89bio Clinical Study Site, Ypsilanti, Michigan
  - 89bio Clinical Study Site, Minneapolis, Minnesota
  - 89bio Clinical Study Site, Rochester, Minnesota
  - 89bio Clinical Study Site, Flowood, Mississippi
  - 89bio Clinical Study Site, Tupelo, Mississippi
  - 89bio Clinical Study Site, St Louis, Missouri
  - 89bio Clinical Study Site, Las Vegas, Nevada
  - 89bio Clinical Study Site, Florham Park, New Jersey
  - 89bio Clinical Study Site, Somers Point, New Jersey
  - 89bio Clinical Study Site, Albuquerque, New Mexico
  - 89bio Clinical Study Site, New York, New York
  - 89bio Clinical Study Site, Asheville, North Carolina
  - 89bio Clinical Study Site, Durham, North Carolina
  - 89bio Clinical Study Site, Fayetteville, North Carolina
  - 89bio Clinical Study Site, Greenville, North Carolina
  - 89bio Clinical Study Site, Winston-Salem, North Carolina
  - 89bio Clinical Study Site, Akron, Ohio
  - 89bio Clinical Study Site, Cincinnati, Ohio
  - 89bio Clinical Study Site, Cleveland, Ohio
  - 89bio Clinical Study Site, Columbus, Ohio
  - 89bio Clinical Study Site, Dayton, Ohio
  - 89bio Clinical Study Site, Liberty Township, Ohio
  - 89bio Clinical Study Site, Westlake, Ohio
  - 89bio Clinical Study Site, Philadelphia, Pennsylvania
  - 89bio Clinical Study Site, Pittsburgh, Pennsylvania
  - 89bio Clinical Study Site, East Greenwich, Rhode Island
  - 89bio Clinical Study Site, Charleston, South Carolina
  - 89bio Clinical Study Site, Columbia, South Carolina
  - 89bio Clinical Study Site, Rapid City, South Dakota
  - 89bio Clinical Study Site, Cordova, Tennessee
  - 89bio Clinical Study Site, Hermitage, Tennessee
  - 89bio Clinical Study Site, Nashville, Tennessee
  - 89bio Clinical Study Site, Austin, Texas
  - 89bio Clinical Study Site, Brownsville, Texas
  - 89bio Clinical Study Site, DeSoto, Texas
  - 89bio Clinical Study Site, Edinburg, Texas
  - 89bio Clinical Study Site, Farmers Branch, Texas
  - 89bio Clinical Study Site, Fort Worth, Texas
  - 89bio Clinical Study Site, Harlingen, Texas
  - 89bio Clinical Study Site, Houston, Texas
  - 89bio Clinical Study Site, Lubbock, Texas
  - 89bio Clinical Study Site, Pearland, Texas
  - 89bio Clinical Study Site, San Antonio, Texas
  - 89bio Clinical Study Site, San Marcos, Texas
  - 89bio Clinical Study Site, Waco, Texas
  - 89bio Clinical Study Site, Sandy City, Utah
  - 89bio Clinical Study Site, West Jordan, Utah
  - 89bio Clinical Study Site, Richmond, Virginia
  - 89bio Clinical Study Site, Seattle, Washington
- Argentina (4):
  - 89bio Clinical Study Site, Buenos Aires
  - 89bio Clinical Study Site, CABA
  - 89bio Clinical Study Site, Capital Federal
  - 89bio Clinical Study Site, Pilar
- Australia (8):
  - 89bio Clinical Study Site, Adelaide
  - 89bio Clinical Study Site, Fitzroy
  - 89bio Clinical Study Site, Greenslopes
  - 89bio Clinical Study Site, Heidelberg
  - 89bio Clinical Study Site, Herston
  - 89bio Clinical Study Site, Murdoch
  - 89bio Clinical Study Site, Perth
  - 89bio Clinical Study Site, South Brisbane
- Belgium (5):
  - 89bio Clinical Study Site, Brussels
  - 89bio Clinical Study Site, Edegem
  - 89bio Clinical Study Site, Genk
  - 89bio Clinical Study Site, Ghent
  - 89bio Clinical Study Site, Roeselare
- Brazil (7):
  - 89bio Clinical Study Site, Barretos
  - 89bio Clinical Study Site, Belo Horizonte
  - 89bio Clinical Study Site, Botucatu
  - 89bio Clinical Study Site, Goiânia
  - 89bio Clinical Study Site, Porto Alegre
  - 89bio Clinical Study Site, Salvador
  - 89bio Clinical Study Site, São José do Rio Preto
- Bulgaria (3):
  - 89bio Clinical Study Site, Gorna Oryahovitsa
  - 89bio Clinical Study Site, Sofia
  - 89bio Clinical Study Site, Stara Zagora
- Canada (7):
  - 89bio Clinical Study Site, Calgary, Alberta
  - 89bio Clinical Study Site, Vancouver, British Columbia
  - 89bio Clinical Study Site, Winnipeg, Manitoba
  - 89bio Clinical Study Site, London, Ontario
  - 89bio Clinical Study Site, Ottawa, Ontario
  - 89bio Clinical Study Site, Toronto, Ontario
  - 89bio Clinical Study Site, Vaughan
- France (13):
  - 89bio Clinical Study Site, Amiens
  - 89bio Clinical Study Site, Dijon
  - 89bio Clinical Study Site, Limoges
  - 89bio Clinical Study Site, Lyon
  - 89bio Clinical Study Site, Montpellier
  - 89bio Clinical Study Site, Nice
  - 89bio Clinical Study Site, Paris
  - 89bio Clinical Study Site, Pessac
  - 89bio Clinical Study Site, Strasbourg
  - 89bio Clinical Study Site, Toulouse
  - 89bio Clinical Study Site, Vandœuvre-lès-Nancy
  - 89bio Clinical Study Site, Vénissieux
  - 89bio Clinical Study Site, Villejuif
- Germany (6):
  - 89bio Clinical Study Site, Chemnitz
  - 89bio Clinical Study Site, Frankfurt
  - 89bio Clinical Study Site, Freiburg im Breisgau
  - 89bio Clinical Study Site, Hanover
  - 89bio Clinical Study Site, Homburg
  - 89bio Clinical Study Site, Münster
- Hong Kong (2):
  - 89bio Clinical Study Site, Hong Kong
  - 89bio Clinical Study Site, Shatin
- 89bio Clinical Study Site, Budapest, Hungary
- Israel (8):
  - 89bio Clinical Study Site, Afula
  - 89bio Clinical Study Site, Beersheba
  - 89bio Clinical Study Site, Haifa
  - 89bio Clinical Study Site, Jerusalem
  - 89bio Clinical Study Site, Nahariya
  - 89bio Clinical Study Site, Petah Tikva
  - 89bio Clinical Study Site, Tel Aviv
  - 89bio Clinical Study Site, Tel Litwinsky
- Italy (9):
  - 89bio Clinical Study Site, Bergamo
  - 89bio Clinical Study Site, Foggia
  - 89bio Clinical Study Site, Milan
  - 89bio Clinical Study Site, Novara
  - 89bio Clinical Study Site, Palermo
  - 89bio Clinical Study Site, Roma
  - 89bio Clinical Study Site, Rome
  - 89bio Clinical Study Site, Rozzano
  - 89bio Clinical Study Site, Torino
- Mexico (7):
  - 89bio Clinical Study Site, Chihuahua City
  - 89bio Clinical Study Site, Cuautitlán Izcalli
  - 89bio Clinical Study Site, Cuernavaca
  - 89bio Clinical Study Site, Jalisco
  - 89bio Clinical Study Site, Mexico City
  - 89bio Clinical Study Site, Mérida
  - 89bio Clinical Study Site, Monterrey
- Netherlands (4):
  - 89bio Clinical Study Site, Amsterdam
  - 89bio Clinical Study Site, Rotterdam
  - 89bio Clinical Study Site, Tilburg
  - 89bio Clinical Study Site, Utrecht
- Poland (6):
  - 89bio Clinical Study Site, Katowice
  - 89bio Clinical Study Site, Krakow
  - 89bio Clinical Study Site, Lodz
  - 89bio Clinical Study Site, Mysłowice
  - 89bio Clinical Study Site, Warsaw
  - 89bio Clinical Study Site, Wroclaw
- 89bio Clinical Study Site, Singapore, Singapore
- South Korea (4):
  - 89bio Clinical Study Site, Bucheon-si
  - 89bio Clinical Study Site, Busan
  - 89bio Clinical Study Site, Daegu
  - 89bio Clinical Study Site, Seoul
- Spain (10):
  - 89bio Clinical Study Site, Almería
  - 89bio Clinical Study Site, Badalona
  - 89bio Clinical Study Site, Barcelona
  - 89bio Clinical Study Site, Córdoba
  - 89bio Clinical Study Site, Madrid
  - 89bio Clinical Study Site, Málaga
  - 89bio Clinical Study Site, Pontevedra
  - 89bio Clinical Study Site, Santander
  - 89bio Clinical Study Site, Santiago de Compostela
  - 89bio Clinical Study Site, Zaragoza
- Taiwan (3):
  - 89bio Clinical Study Site, Chiayi City
  - 89bio Clinical Study Site, Kaohsiung City
  - 89bio Clinical Study Site, Tainan
- Turkey (Türkiye) (5):
  - 89bio Clinical Study Site, Bornova, İzmir
  - 89bio Clinical Study Site, Merkez, Rize Province
  - 89bio Clinical Study Site, Ankara
  - 89bio Clinical Study Site, Istanbul
  - 89bio Clinical Study Site, Yüreğir
- United Kingdom (9):
  - 89bio Clinical Study Site, Aberdeen
  - 89bio Clinical Study Site, Bristol
  - 89bio Clinical Study Site, Hants
  - 89bio Clinical Study Site, Leeds
  - 89bio Clinical Study Site, London
  - 89bio Clinical Study Site, Oxford
  - 89bio Clinical Study Site, Plymouth
  - 89bio Clinical Study Site, Port Talbot
  - 89bio Clinical Study Site, Southampton